CLINICAL TRIAL: NCT07326202
Title: Gait Asymmetry And Its Relationship With Neck Pain And Muscles Strength In Patients With Cervical Radiculopathy
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hossam Abdel Wahab Mohamed, Principal investigator, Cairo University
Other Study IDs: P.T.REC/012/005942
Record Dates: First submitted 2025-12-24; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Cervical Radiculopathy
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cervical radiculopathy group: Sixty-one patients with cervical radiculopathy of both sexes will participate in this study. Patients will be diagnosed as having cervical radiculopathy by neurologist based on a careful clinical examination and will be confirmed by investigations as magnetic resonance imaging (MRI).

INTERVENTIONS:
Other:

SUMMARY:
This study will be conducted to:

* Investigate the relationship between neck pain severity and bilateral gait symmetry in patients with cervical radiculopathy.
* Investigate the relationship between deep neck flexors strength and gait symmetry in patients with cervical radiculopathy.
* Investigate the relationship between upper limb muscles strength and bilateral gait symmetry in patients with cervical radiculopathy.
* Determine factors predicting bilateral gait asymmetry in patients with cervical radiculopathy.

DETAILED DESCRIPTION:
Cervical pain and upper limb radiculopathy put a huge burden on patients due to its sensory dysfunction manifestations and also affect its motor capabilities, specifically the gait performance, understanding how cervical and upper limb pain or/and weakness contribute to gait disturbance can guide us to make a better assessment and rehabilitation program for each patient individually.

Gait symmetry is considered as a very important factor to guarantee a safe and effective walking and for the daily movement, recent studies found out that patients with chronic neck pain and radiculopathy have slower gait pattern and increase of gait asymmetry which can impair balance and functional mobility. Also, the alteration of the cervical and upper limb muscle strength can impair the whole-body dynamic stability and increase the gait asymmetry.

Altered gait symmetry has been linked to increase the risk of falling and disability, so getting to know some of its contributors and treat it (such as specific muscle strengthening) can enhance patient mobility and reduce fall morbidity.

To our best knowledge, there are no studies about the relationship between neck pain, muscle strength in patients with cervical radiculopathy, so this study will be conducted to investigate the gait asymmetry and its relationship with neck pain and muscles strength in patients with cervical radiculopathy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unilateral cervical radiculopathy at level of C5-C6 and C6-C7 confirmed by MRI.
* Patient's age will be ranged from 40 to 50 years.
* Patients with chronic symptoms > 3 months.
* Patients with decreased strength in cervical or upper limb muscles.
* Ability to walk independently without assistive devices.
* Patients with normal body mass index (BMI) (< 30kg/m²) .

Exclusion Criteria:

* Bilateral cervical radiculopathy.
* History of cervical spine surgery or instability.
* Diagnosed with myelopathy, canal stenosis, or severe disc protrusion.
* History of vestibular dysfunction, stroke, or severe cognitive impairment.
* Any Lower limb dysfunction affecting walking.
* Peripheral neuropathy or uncontrolled diabetes.
* Psychiatric diseases
* Pregnancy.

Ages: 40 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Sixty one patients with cervical radiculopathy of both sexes will participate in this study. Patients will be diagnosed as having cervical radiculopathy by neurologist based on a careful clinical examination and will be confirmed by investigations as magnetic resonance imaging (MRI). Patients will be selected from the Outpatient Clinic of Faculty of Physical Therapy, and the British University in Egypt
Sampling Method: Non-Probability Sample
Enrollment: 61 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-03-25 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Pain Assessment | 1 day
  The level of upper limb and neck pain will be captured separately with the Numeric Pain Rating Scale (NPRS). Using an 11-point scale, ranging from 0 (no pain) to 10 (worst pain imaginable), participants will be asked to answer the following question: "On a scale of 0 to 10, where 0 = no pain and 10 = worst pain, evaluate the intensity of your neck pain at this moment ". The same question will be asked for the upper limb. The NPRS is frequently used in clinical studies in association with the neck disability index.
Assessment of function and disability | 1 day
  Arabic version of Neck Disability Index (NDI) will be used to assess disability and function limitation caused by neck pain. It has demonstrated excellent internal consistency (Cronbach's alpha between 0.88 and 0.94) and test-retest reliability (ICC = 0.90-0.98). It includes 10 items, each scored on a 0-5 scale, about: personal care, lifting, reading, concentration, work, driving, and sleeping. The total maximum score is 50 and categorize disability from none to complete , The Arabic version of NDI is a strong valid method for assessing self-rated disability in patients with neck pain with excellent "test-retest" reliability. Based on the total score (out of 50), disability will be categorized as:
  0-4 = no disability, 5-14 = mild, 15-24 = moderate, 25-34 = severe, >34 = complete disability
strength of deep neck flexors | 1 day
  Pressure Biofeedback Unit (PBU) will be used to assess deep neck flexor strength.
  From a supine position and both knees bent in flexion and arms relaxed at the sides. The PBU cuff will be placed under the suboccipital region of his neck and then inflated to a baseline pressure of 20 mmHg. Patients will be instructed to perform a gentle chin in motion without lifting their heads off the surface or activating superficial muscles. The patient will then be guided to increase the pressure in 2 mmHg stages to a maximum of 30 mmHg, and to hold each stage for 10 seconds taking no rest intervals between his attempts. The maximum pressure which he achieves and holds correctly without compensatory strategies will be recorded. 3 trials will be conducted.
Upper limb strength assessment | 1 day
  Upper limb strength will be measured using a hand-held dynamometer. Participants will be seated in upright posture, with their shoulders adducted and neutrally rotated, and their elbows will be flexed at 90 degrees, their forearms will be placed in a neutral position, and their wrists extended between 0-30 degrees, testing protocol. Each participant will be instructed to grip the dynamometer with his maximum effort for about 3-5 seconds. The participant will receive consistent verbal encouragement from the assessor to ensure maximal voluntary contraction is achieved. Each participant will perform 3 trials on their affected side, with a one-minute rest between his attempts to avoid muscle fatigue.
Cadence | 1 day
  The Tekscan Strideway™ system will be used to objectively assess spatiotemporal gait parameters for all participants with cervical radiculopathy. Cadence is the number of steps taken per minute (steps/minutes).
Gait Velocity | 1 day
  The Tekscan Strideway™ system will be used to objectively assess spatiotemporal gait parameters for all participants with cervical radiculopathy. Gait Velocity is the average walking speed, calculated as Gait Distance divided by Gait Time (centimeter/second).
Symmetry Index (SI) | 1 day
  The Tekscan Strideway™ system will be used to objectively assess spatiotemporal gait parameters for all participants with cervical radiculopathy. Symmetry Index (SI) is a calculated percentage representing the degree of asymmetry between the right and left sides for any given gait parameter (%).
  Formula used:
  SI = [(Right - Left) / 0.5 * (Right + Left)] * 100.
Step Time symmetry index | 1 day
  The Tekscan Strideway™ system will be used to objectively assess spatiotemporal gait parameters for all participants with cervical radiculopathy. Step time is the percentage of asymmetry between the right step time and the left step time (%).
Step Length symmetry index | 1 day
  The Tekscan Strideway™ system will be used to objectively assess spatiotemporal gait parameters for all participants with cervical radiculopathy. Step Length is a percentage of asymmetry between the right step length and the left step length (%).
Single Support Time symmetry index | 1 day
  The Tekscan Strideway™ system will be used to objectively assess spatiotemporal gait parameters for all participants with cervical radiculopathy. Single Support Time is the percentage of asymmetry between the average right single support time and the average left single support time (%).
Double Support Time symmetry index | 1 day
  The Tekscan Strideway™ system will be used to objectively assess spatiotemporal gait parameters for all participants with cervical radiculopathy. Double Support Time is the percentage of asymmetry between the average right total double support time and the average left total double support time (%).

CONTACTS AND LOCATIONS:
Overall Officials: Ebtesam Fahmy, Professor, Study Director — Cairo University; Nagwa Rehab, Professor, Study Chair — Cairo University
Locations (1):
- Hossam Abdelwahab mohamed, Cairo, Egypt